CLINICAL TRIAL: NCT01724593
Title: Functional Recovery in Critically Ill Children - the Wee-Cover Pilot Study
Brief Title: Functional Recovery in Critically Ill Children
Status: Completed | Type: Observational
Sponsor: Karen Choong (Other)
Responsible Party: Sponsor-Investigator, Karen Choong, Associate Professor, McMaster University
Organization: McMaster University (Other)
Other Study IDs: HHS REB No. 12-475
Record Dates: First submitted 2012-10-30; First posted 2012-11-12 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Critical Illness; Children
Keywords: functional recovery, critical illness, pediatrics
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Cohort: No Intervention

SUMMARY:
Intensive Care Unit-acquired weakness (ICU-AW) is a well-recognized, important and preventable sequelae of critical illness, affecting up to 60% of adult ICU patient. ICU-AW is associated with increased mortality and length of stay, and negatively impacts long-term functional outcomes and quality of life in affected patients and their caregivers. While delayed mobilization adversely affects clinical outcomes, early rehabilitation in the critically ill adult population is safe, feasible, cost effective, results in more ventilator free-days and better functional outcomes at hospital discharge. In contrast, there is a paucity of this research in pediatrics. Our research suggests that immobilization is common in critically ill children, and rehabilitation is delayed particularly in the sickest children who are arguably at highest risk of morbidity. It is unclear however, whether delayed rehabilitation leads to adverse outcomes in critically ill children, as has been demonstrated in adults. Our objectives of this study are to evaluate if immobilization and delayed rehabilitation negatively impacts short-term clinical outcomes and the time to functional recovery in critically ill children. The investigators hypothesize that the following factors may influence functional recovery and morbidity in critically ill children:

* Pre-morbid condition
* Age
* Time-to-initiation of acute rehabilitation
* Critical illness disease severity

DETAILED DESCRIPTION:
Overall Study objectives:

1. To describe the functional recovery following prolonged immobility and delayed rehabilitation in critically ill children.
2. To explore the predictors of impaired functional recovery following immobilization in critically ill children.

Prior to conducting a definitive multi-centre study to answer our research questions and achieve our study objectives above, we will conduct a pilot study in order to demonstrate feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age over 12 months to 17 years
* PCCU stay of ≥ 48 hours
* Patient is limited to bed-rest and has not been mobilized during the first 48 hours of PCCU admission
* Equal to or greater than one organ dysfunction on PCCU admission (as measured by PELOD)
* Informed consent of patient/substitute decision maker.

Exclusion Criteria:

* Age: < 12 months or ≥18 years
* Patients admitted to step-down/intermediate care
* Patients transferred from Neonatal intensive care unit and never discharge home.

iv) Patients who are already mobilizing well, or are at baseline functional status at time of screening v) Admission diagnosis of a neuromuscular disorder: e.g. Acute Guillain-Barré Syndrome, Botulism, Myasthenia Gravis), or acute spinal cord injury/transverse myelitis vi) Not expected to survive PCCU/hospital stay vii) Previously enrolled into study less than 6 months ago and/or still undergoing study procedures at time of screening

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically Ill Children
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Feasibility | 12 months
  Feasibility will be determined by the consent and enrolment rate, and the protocol adherence and follow-up rates.

SECONDARY OUTCOMES:
Functional Recovery | Baseline, 3 and 6 month follow-up
  Functional Recovery will be measured by the following standardized, validate pediatric assessment tools of function, as defined by the International Classification of Functioning, Disability and Health (ICF): 1) Pediatric Evaluation of Disability Inventory (PEDI); 2) Participation and Environment Measure - children and youth version (PEM-CY), and preschool version; 3) Pediatric Overall Performance Category score (POPC); 4) Pediatric Cerebral Performance Category Score (PCPC)
Pediatric Critical care Unit (PCCU) clinical outcomes | at 30 days and duration of hospitalization
  PCCU outcomes will be assessed by the following: Ventilator-free days, PCCU mortality, length of PCCU and hospital stay, and the incidence of PCCU-acquired weakness
Muscle Strength | Hospital discharge and at 3 and 6 month follow-up
  In an age-appropriate subgroup, the following measurements will be conducted:
  * Muscle Strength and aerobic fitness testing (age ≥ 5 years, and/or able to cognitively and physically comply with strength and fitness tests)
  * Measurement of muscle strength using BIODEX and hand grip strength, and assessment of lean mass (Bioelectrical impedance analysis)
Parental or caregiver stress | 3 month follow-up
  Parental or caregiver stress will be measured with the Parental Stress Index (PSI)

OTHER OUTCOMES:
Feasibility and reliability of screening for PCCU-acquired weakness | Duration of Hospitalization, 3 and 6 months follow-up
  The most appropriate method of screening and diagnosing PCCU-acquired weakness has not been well established given the many challenges in ascertainment in this population. Hence, one of the objectives of this study is to determine whether manual muscle strength testing is a feasible and reliable method of screening for this important disorder in the critically ill pediatric population. Muscle strength will be quantified clinically using the (MRC) score by 2 independent assessors. For a subset of age appropriate (≥ 4 years), we will determine their hand-grip strength using a hand dynamometer or Martin Vigorimeter, depending on their age.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MB, BCh, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada